CLINICAL TRIAL: NCT02675374
Title: Hemodynamic Instability Prevented With Polaramine® Infusion Before Extracorporeal Circulation
Acronym: HIPPIE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHUBX 2014/13
Record Dates: First submitted 2016-01-11; First posted 2016-02-05 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Hemodynamic Instability; Vasoplegic Syndrome
Keywords: Cardiac surgery; cardiopulmonary bypass; dexchlorpheniramine; H1 blockers; norepinephrine; histamine release
MeSH Terms: conditions — Vasoplegia | interventions — dexchlorpheniramine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 24 patients
  Interventions: Drug: dexchlorpheniramine (Polaramine®) injection
- Control group (Placebo Comparator): 24 patients
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: dexchlorpheniramine (Polaramine®) injection — 5 minutes before CPB, patients will receive 10 mg (2 ml) of Polaramine®
  Arms: Treatment group
Drug: Placebo injection — 5 minutes before CPB, patients will receive 2 ml of normal saline
  Arms: Control group

SUMMARY:
This single-institution randomized controlled trial prospective will enrolled 48 patients scheduled for an aortic valve replacement. The objective of the present investigation is to determine the role of Polaramine® on reducing hemodynamic instability after separation from cardiopulmonary bypass (CPB) during cardiac surgery. Our hypothesis is that Polaramine® play an important role reducing dysfunction of the autonomic nervous system and hemodynamic stability after separation from CPB.

DETAILED DESCRIPTION:
Vasoplegic syndrome is recognized as a common complication after CPB. Its incidence ranges from 5% to 25% after cardiac surgery requiring CPB. Such syndrome is related to an inflammatory reaction, which is attributed to the CPB. This syndrome is typically characterized by a combination of different parameters with low specificity and sensitivity, such as low systemic vascular resistance leading to a hypotension imposing perfusion of vasopressors with high or normal cardiac outputs.

Investigators preliminary data suggest that vasoplegic syndrome might be related to heart manipulation during surgery. Tearing maneuvers performed on the heart chambers trigger peaks pressure stimulating, consequently, baroreceptors and finally resulting in arteriovenous vasodilation via neurogenic and endogenous pathways. According to investigators initial investigation, such reaction appears to be related to basophils degranulation and release of vasoactive substances.

The hypothesis of the present trial is that a reduction of basophils degranulation and release of vasoactive substances via an antihistaminic could lower the incidence of the vasoplegic syndrome. This study aims to determine the effect of an antihistamine (dexchlorpheniramine (Polaramine®)) administered intravenously before CPB, on the vasoplegic syndrome incidence after separation from CPB.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 and older
* Post menopausal women
* Patients scheduled for an aortic valve replacement with a traditional sternotomy and CPB

Exclusion Criteria:

* Patients with a left ventricular ejection fraction lower than 40%
* Patients with pulmonary arterial hypertension higher than 50mm of Hg,
* Redo cardiac surgery,
* Atrioventricular and intraventricular conduction disturbances
* Epilepsy or convulsions
* Atopic disease
* Women of childbearing potential
* Patients at risk of glaucoma
* Patients with therapy interacting with dexchlorpheniramine (Polaramine®).
* Patients unable to provide a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-05 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Assesment of patients proportion with abnormal ratio of sympathic-parasympathetic balance (>1.2) | Day 0
  The calculation of every ratio will be made by a software in the department
Assesment of patients proportion with abnormal ratio of sympathic-parasympathetic balance (>1.2) | Day 1
  The calculation of every ratio will be made by a software in the department
Assesment of patients proportion with abnormal ratio of sympathic-parasympathetic balance (>1.2) | Day 2
  The calculation of every ratio will be made by a software in the department

SECONDARY OUTCOMES:
Blood dosage of histamine | Day 0
Immunophenotypage of basophilic polynuclears | Day 0
Peaks of pressure measure in the lung artery perioperative | Day 0, day 1, day 2
Assesment of the postoperative complications incidence | Day 28, month 6
Measure of the amount of fluids delivered | Day 0, day1, day 2
Measure of the amount of catecholamine infused | Day 0, day 1, day 2
Duration of hospital stay | Day 28
Mortality | Day 28, month 6
Collection of adverse events potentially related to the treatment | Day 0, day1, day 2, day 28, month 6
Assesment of patients proportion presenting metabolic disease, with abnormal ratio of sympathic-parasympathetic balance (>1.2) | Day 0, day 1, day 2

CONTACTS AND LOCATIONS:
Overall Officials: Cédrick ZAOUTER, Dr, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France